CLINICAL TRIAL: NCT05466994
Title: A Phase II Randomized Controlled Trial to Determine the Efficacy of an auGmented reAlity gaMe in pediatrIc caNcer Patients Who Are Opioid Naïve Undergoing Surgery to Reduce Postoperative Opioid Use (GAMING-ON Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0336; NCI-2022-05979 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pediatric ALL; Cancer
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1(Spellbound) (Other): Participants will play the game using the iPad's standard camera, which will show you your hospital room and the decals as they appear in the real world.
  Interventions: Other: IPAD
- Group 2 (Spellbound) (Other): Participants will play the game using augmented reality
  Interventions: Other: Augmented Reality

INTERVENTIONS:
Other: IPAD — Participant will play a game through (standard camera) participants will be able to the hospital room and decals as they appear in the real world
  Arms: Group 1(Spellbound)
Other: Augmented Reality — Participants will play a game through (devices camera and application) let us participants view the real world
  Arms: Group 2 (Spellbound)

SUMMARY:
To learn if playing an augmented reality game called SpellBound can reduce pain and the need for opioids in young patients scheduled for surgery.

DETAILED DESCRIPTION:
Primary Objective:

•To assess the efficacy of SpellBound's AR-enabled scavenger hunt to reduce the rate of 90-day opioid use in pediatric cancer patients undergoing surgery compared to a control non-AR game in a randomized controlled trial.

Secondary Objectives:

To assess the effect of AR versus non-AR control technology in pediatric oncology patients, including:

* Inpatient opioid use
* Average daily inpatient pain score
* Number of opioid requests during the hospital stay
* Inpatient PedsQL (quality of life) questionnaire score
* Ambulation/"out of bed" movement
* Number days to discharge-ready status
* Patient experience assessed by satisfaction scores on a questionnaire designed by MD Anderson Cancer Center Child Life team.
* Outpatient opioid consumption reported at 30, 60, and 90 days
* Outpatient pain scores reported at 30, 60, and 90 days
* Outpatient PedsQL scores reported at 30, 60, and 90 days
* Potential adverse events related to the use of AR (i.e., falls).

ELIGIBILITY:
Inclusion Criteria:

1. Ages 5-15
2. English and Spanish-speaking parents/legal guardians and patients
3. Undergoing major surgery for cancer requiring postoperative hospitalization is defined as ≥2 hours of duration of surgery and requiring postoperative hospital admission of at least one night
4. Expected to be prescribed postoperative inpatient opioids
5. Have never taken opioids or have had no daily opioid use within the last 30 days before surgery
6. Sufficient cognitive capacity to comprehend and interact with the game. This is defined as the ability to utilize mobile technology (use iPad with or without assistance) and activate and respond to AR experiences within the app as determined by the clinician.
7. Both the child and a legal guardian are willing and able to provide informed consent.

   * The range from 5-to 15 is based on a recent pilot RCT in which the PI found that older adolescents (>15 years of age) were disinterested in the interactive game.

Exclusion Criteria:

1. Patients with any daily opioid use within 30 days before surgery.
2. History of documented peripheral neuropathy secondary to cancer treatment
3. Inability to demonstrate an understanding of the game from English instructions
4. Any additional concerns based on the study physicians' assessments

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2026-01-13 (Actual); Study Completion 2026-01-13 (Actual)

PRIMARY OUTCOMES:
Pediatric Quality of Life Inventory Questionnaires | through completion of study, an average of 1 year
  Quality of life assessment-Age-appropriate Pediatric Quality of Life Inventory (PedsQL)29 paper surveys will be administered to the patient (self-report) or guardian (proxy) when patients reach discharge-ready status. Score scales (0-4) 0-Never/4 Almost Always

CONTACTS AND LOCATIONS:
Overall Officials: Juan Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - M D Anderson Cancer Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT05466994/ICF_000.pdf